CLINICAL TRIAL: NCT03611244
Title: Prevention of Scoliosis in Patients With Duchenne Muscular Dystrophy Using Portable Seat Device Devised to Maintain Lumbar Lordosis : 5 Year Follow up Study
Brief Title: Prevention of Scoliosis in Patients With Duchenne Muscular Dystrophy Using Portable Seat Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyung-ik Shin, Associate professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1806-171-955 SNUH
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Scoliosis Neuromuscular; Duchenne Muscular Dystrophy; Lordosis Lumbar
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): When loss of ambulation was observed in patients with Duchenne muscular dystrophy, portable seat device devised to maintain lumbar lordosis were applied within 1 year, and then compliance with the the device were evaluated at 6-month intervals for 5 years.
  Interventions: Device: Portable seat device devised to maintain lumbar lordosis
- Control group (No Intervention): Analysis of retrospective medical records who had not been applied portable seat device devised to maintain lumbar lordosis

INTERVENTIONS:
Device: Portable seat device devised to maintain lumbar lordosis — The posterior lumbar spine pads are used to maintain lumbar lordosis and fix it with the shoulder strap so that the hip does not slip forward (so that it does not become a sacral sitting posture).
  The seat is equipped with a 5 cm air filled villus cushion to relieve pressure on the ischial tuberosity when sitting for a long time. The portable seat device can be moved so that the DMD can sit on the device even when sitting in a wheelchair or a chair for home, school, or outdoors, so that the lumbar lordosis can be constantly maintained.
  Arms: Experimental group

SUMMARY:
This study will be conducted without blind method. The portable seat device devised to maintain lumbar lordosis will be made within 1 year after the loss of ambulation in the participants with Duchenne muscular dystrophy with prospective design.

In the control group, the presence of scoliosis will be calculated 5 years after the loss of ambulation in participants with Duchenne muscular dystrophy through analysis of retrospective medical records who had not been applied the portable seat device.

DETAILED DESCRIPTION:
In the retrospective data of Seoul National University Children's Hospital, the incidence of 5-year scoliosis in the control group in the past using steroids alone was 70% in patients with confirmed Duchenne muscular dystrophy. When applying the portable seat device (experimental group), the incidence of scoliosis is expected to decrease to 50% (ie, 35% because of 50% of 70%) compared with using steroid alone.

In this study, investigators will enroll 70 control subjects who did not use the portable seat device through retrospective data. The number of subjects required to show the difference between the significance level of 5% and the power of 80% was 19, and 28 participants with DMD are required considering 30% dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Duchenne muscular dystrophy diagnosed by genetic study were included.

  1. Within 1 year after loss of ambulation (Vignos scale 7 points or more)
  2. Condition without scoliosis
  3. Conditions that do not have physical (eg, cerebral palsy) and mental (eg, moderate or higher intellectual disability) comorbid conditions that will affect the use of postural seat device.

Exclusion Criteria:

1. Patients who do not agree to participate in this study
2. Patients not taking steroids
3. Patient with scoliosis

Ages: 7 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of scoliosis | 5 years after loss of ambulation
  Frequency of scoliosis more than 10 degrees on spine x-ray on supine position

SECONDARY OUTCOMES:
Incidence of scoliosis | "Day 0", "Month 6" "Month 12" "Month 18" "Month 24" "Month 30" "Month 36" "Month 42" "Month 48" "Month 54" "Month 60"
  Comparison of cobb's angle on spine x-ray on supine position

CONTACTS AND LOCATIONS:
Overall Officials: You Gyoung Yi, M.D., MSc, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No